CLINICAL TRIAL: NCT04764227
Title: Phase II Study of Postoperative Concurrent Chemoradiotherapy for Esophageal Squamous Cell Carcinoma (ESO- Shanghai 17)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Prof, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO- Shanghai 17
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Esophagus Cancer; Esophageal Squamous Cell Carcinoma; Chemoradiotherapy; Radiation Therapy; Postoperative
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent chemoradiotherapy group (Experimental): Interventions:
  * Chemotherapy: Paclitaxel 50mg/m2/d, ivgtt over 3 hours, d1; Carboplatin AUC=2, ivgtt, d1; qw*5
  * Radiotherapy: A total dose of 50.4Gy will be delivered in 28 fractions at 1.8Gy/fraction, 5 fractions per week in 6 weeks. The CTV encompassed the bilateral supraclavicular, superior mediastinal, and subcarinal regions.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — paclitaxel 50mg/m2/d, ivgtt over 3 hours, d1, qw*5
Drug: Carboplatin — carboplatin AUC=2, ivgtt, d1, qw*5
Radiation: Radiotherapy — 1.8Gy/d, d1-5/week, 28Fx

SUMMARY:
The purpose of this study is to evaluate safety and 2-year local control rate for postoperative concurrent chemoradiotherapy for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age 18-75;
* ECOG 0-2;
* Esophageal squamous cell carcinoma, radical surgery ≤ 3 months, R0 resection;
* The operative incision healed well;
* T3-4N0M0, T1-4N1-3M0 (according to AJCC2009);
* No radiotherapy, chemotherapy or other treatments pre (post) surgery;
* PS ECOG 0-2;
* Life expectancy of more than 3 months;
* Hemoglobin (Hb) ≥ 9 g/dL, WBC ≥ 3 x 109/L, Neutrophils (ANC ) ≥ 1.5 x 109/L, Platelet count (Pt) ≥ 100 x 109/L;
* Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL< 1.5 x ULN;
* Renal function: creatinine < 1.5 x ULN
* No immuno-deficiency;
* Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

* Complete esophageal obstruction after surgery, Esophageal perforation, Haematemesis;
* Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years;
* Participation in other interventional clinical trials within 30 days;
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives;
* Drug addiction, Alcoholism or AIDS;
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior;
* Unsuitable to be enrolled in the trial in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 2 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Shen J, Ai D, Chen Y, Liu Q, Deng J, Hao S, Zhang X, Zhang J, Zhang Y, Chu L, Sun Y, Zhang Y, Xiang J, Miao L, Chen H, Zhu H, Zhao K. Postoperative chemoradiotherapy for esophageal squamous cell Carcinoma: Results from ESO-Shanghai 17 and joint analyses for phase II clinical trials. Clin Transl Radiat Oncol. 2025 Nov 21;57:101073. doi: 10.1016/j.ctro.2025.101073. eCollection 2026 Mar. PMID 41531940